CLINICAL TRIAL: NCT05800041
Title: A Exploratory Trial to Evaluate the Safety, Tolerability, Pharmacokinetics (PK), Pharmacodynamics (PD), Immunogenicity, and Preliminary Efficacy of WTX221 Infusion in Patients With Refractory Gout
Brief Title: A Exploratory Trial of WTX221 in Refractory Gout Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Westlake Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Evolve-101
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Gout Tophus
MeSH Terms: interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Treatment group A (Experimental): WTX221 low dose
  Interventions: Drug: WTX221
- Treatment group B (Experimental): WTX221middle dose
  Interventions: Drug: WTX221
- Treatment group C (Experimental): WTX221 high dose
  Interventions: Drug: WTX221

INTERVENTIONS:
Drug: WTX221 — Drug: WTX221 WTX221 infusion once every 30 days for two doses in total Drug: CTX Co-administration of CTX and WTX221 at the initial infusion
  Other Names: cyclophosphamide

SUMMARY:
This trial is a single-center, open-label designed investigator-initiated clinical study (IIT) to investigate the safety, tolerability, PK, PD, immunogenicity, and preliminary efficacy of multiple doses of WTX221 infusion combined with a single dose of the immunosuppressive agent cyclophosphamide (CTX) to induce immune tolerance.

The trial consisted of a Screening Period (14 days), a First Dose Period (30 days), a Second Dose Period (30 days), and a Safety Follow-up Period (150 days) for a total of 224 days.

DETAILED DESCRIPTION:
Refractory gout is usually associated with persistently swollen and tender joints, chronic pain, reduced functional status, impaired quality of life, and joint destruction，most of the patients can't tolerate urate-lowering therapy(ULT)or receive adequate dose of ULT treatment recommended to control Serum uric acid (SUA) to target level.

WTX221 is designed to induce antigen-specific immune tolerance. WTX221 is made of urate oxidase(UOX) molecules conjugated on the surface of Red blood cells(RBCs), which can induce antigen-specific immune tolerance to UOX in vivo by making use of it's natural biologic characteristics. WTX221 infusion combined with a single dose CTX to induce immune tolerance.

The trial consisted of a Screening Period (14 days), a First Dose Period (30 days), a Second Dose Period (30 days), and a Safety Follow-up Period (150 days) for a total of 224 days.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand the purpose and requirements of this trial, voluntarily participate in the clinical trial and sign the informed consent form, and be able to complete all trial processes as required by the protocol;
* Subject is ≥ 18 years of age;
* Patients with refractory gout: multiple tophi, more than 2 sites;
* Subjects (males and females) must agree to be free of childbearing potential and willing to use effective contraception with their partner and have no plans to donate sperm or eggs during the trial and for at least 1 year after the infusion.

Exclusion Criteria:

* Patients with allergic diseases or specific allergic history, or possible allergic to the study drug and any of its components or related preparations;
* Patients unable to communicate or cooperate with medical staff due to neurological, mental illness or language disorder, which affects patient compliance;
* Having any past or present medical history that may affect the safety of the trial or the in vivo process of the drug, especially history of cardiovascular, liver, kidney, digestive tract, lung, spleen, nerve, blood, tumor, immune or metabolic disorders that are considered clinically significant by the investigator;
* Participated in other drug or medical device clinical trials within 3 months before screening;
* Patients who have received intravenous anti-infective treatment or active infection within 14 days before administration;
* Patients with history of allogeneic organ, bone marrow transplantation or stem cell transplantation;
* Patients with laboratory abnormalities that are clinically significant:
* The investigator believes that it will prevent the subject from following and completing any other circumstances of the study protocol;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2023-04-10 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of multiple doses of WTX221 infusion combined with a single dose of cyclophosphamide in patients with refractory gout. | from the first WTX221 infusion to 210 days
  Adverse Events and Serious Adverse Events

SECONDARY OUTCOMES:
To evaluate the pharmacokinetic (PK) profile of multiple doses of WTX221 infusion combined with a single dose of cyclophosphamide in patients with refractory gout; | from the first WTX221 infusion to 210 days
  Functional protein content in blood (PK)
To evaluate the pharmacodynamic (PD) profile of multiple doses of WTX221 infusion combined with a single dose of cyclophosphamide in patients with refractory gout | from the first WTX221 infusion to 210 days
  plasma uric acid(UA) level
To evaluate the preliminary efficacy of multiple doses of WTX221 infusion combined with a single dose of cyclophosphamide in patients with refractory gout | from the first WTX221 infusion to 60days Number of gout flares in subjects (within 60 days);
  plasma UA level < 360 umol/L
To evaluate immunogenicity (ADA) levels of multiple doses of WTX221 infusion combined with a single dose of cyclophosphamide in patients with refractory gout | from the first WTX221 infusion to 210days
  ADA incidence rate

IPD SHARING:
Plan to Share IPD: No